CLINICAL TRIAL: NCT04418336
Title: Endoscopic Pilonidal Sinus Treatment (EPSIT) Versus Sinus Laser Closure (SiLaC) Versus Lay Open Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.19.04.495.R1 - 2019/05/12
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endoscopic Pilonidal sinus treatment (EPSIT) (Active Comparator): Endoscopic Pilonidal sinus treatment (EPSIT)
  Interventions: Procedure: Endoscopic Pilonidal sinus treatment (EPSIT) versus Sinus Laser Closure (SiLaC) versus lay open technique
- Sinus Laser Closure (SiLaC) (Active Comparator): Sinus Laser Closure (SiLaC)
  Interventions: Procedure: Endoscopic Pilonidal sinus treatment (EPSIT) versus Sinus Laser Closure (SiLaC) versus lay open technique
- lay open technique (Active Comparator): lay open technique
  Interventions: Procedure: Endoscopic Pilonidal sinus treatment (EPSIT) versus Sinus Laser Closure (SiLaC) versus lay open technique

INTERVENTIONS:
Procedure: Endoscopic Pilonidal sinus treatment (EPSIT) versus Sinus Laser Closure (SiLaC) versus lay open technique — Endoscopic Pilonidal sinus treatment (EPSIT) versus Sinus Laser Closure (SiLaC) versus lay open technique in sacrococcygeal Pilonidal sinus treatment

SUMMARY:
Aim of the work To compare Sinus Laser closure versus lay open technique versus Endoscopic pilonidal sinus treatment as regards recurrence rate, operative data, postoperative pain, intra and postoperative complications, healing time and return to daily activity.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptoms from sacrococcygeal pilonidal sinus .

Exclusion Criteria:

* Abscess formation
* Immunodeficiency.
* Patients with congenital asymptomatic pits.
* Patient with psychiatric disease disabling surgical intervention. . Pregnant females.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence | one year
  Recurrence of pilonidal sinus after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt